CLINICAL TRIAL: NCT06206603
Title: Epigenetic Regulation of Colorectal Polyps and Cancer and Its Traceability in Blood
Brief Title: Epigenetic Regulation of Colorectal Polyps and Cancer
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: EPIPOL
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Colorectal Polyp; Colorectal Adenoma; Colorectal Neoplasms
Keywords: Colorectal cancer; Colorectal polyps
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Colorectal polyps: Biopsies will be obtained from the polyp and from adjacent healthy intestinal mucosa. A blood sample will be collected to investigate if certain microRNA/mRNA profiles are traceable in the blood.
  Interventions: Diagnostic Test: Intestinal biopsies; Diagnostic Test: Blood sample
- Colorectal cancer: Biopsies will be obtained from the cancer and from adjacent healthy intestinal mucosa. A blood sample will be collected to investigate if certain microRNA/mRNA profiles are traceable in the blood.
  Interventions: Diagnostic Test: Intestinal biopsies; Diagnostic Test: Blood sample
- Healthy controls: Biopsies will be obtained from predefined locations in the colon and rectum. A blood sample will be collected to investigate if certain microRNA/mRNA profiles are traceable in the blood.
  Interventions: Diagnostic Test: Intestinal biopsies; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Intestinal biopsies — Approximately 6 biopsies (each around 2-3mm in size) are taken from the polyp or cancer, as well as adjacent healthy intestinal mucosa, during a scheduled colonoscopy. For healthy controls, around 6 biopsies are taken from the healthy intestinal mucosa. The intestinal biopsies are frozen at -80 degrees Celsius.
Diagnostic Test: Blood sample — A venous blood sample (10ml) will be taken in connection with the colonoscopy. Patients typically receive an intravenous needle for the administration of sedatives and pain-relieving medications during the colonoscopy, so the current blood sample does not cause any additional needle sticks or discomfort for the patient. The blood sample is centrifuged, and the plasma is frozen at -80 degrees Celsius.

SUMMARY:
The goal of this study is to learn about the epigenetic and genetic regulation (microRNA/mRNA) of colorectal polyps and their evolvement as polyps and to colorectal cancer. Furthermore, the study aims at investigating whether certain epigenetic features, linked to polyps and/or cancer are traceable in blood samples.

The main questions the study aims to answer are:

1. Are there specific microRNA/mRNA that are expressed in different types of polyps and cancers and their respective stages?
2. Is microRNA/mRNA expression in polyps and cancer traceable in blood from the same patient?
3. Is the intestinal microbiata correlated with colorectal polyps and cancer and their microRNA/mRNA expression?

Type of study: clinical trial Participant population Participants consist of patients undergoing a scheduled colonoscopy where a polyp or cancer is discovered. Healthy controls, with normal colonoscopy findings will be enrolled.

Biopsies will be obtained from polyps/cancers and from normal surrounding intestinal mucosa. Biopsies will be obtained from defined intestinal locations from healthy controls. Blood samples will be collected from all participants.

Researchers will compare microRNA/mRNA and microbiota in patients with polyps/cancers and their respective stages as well as healthy controls. Comparisons include biopsies and blood samples.

DETAILED DESCRIPTION:
Scientific Question The study aims to investigate the epigenetic regulation of polyps in the colon and rectum in patients undergoing colonoscopy. The intention is to examine the expression of microRNA/mRNA in blood and intestinal tissue in patients with colorectal polyps or colorectal cancer, as well as in healthy controls. The goal is to learn more about microRNA/mRNA alterations responsible for the evolvement of colorectal polyps and cancer as well as to trace specific microRNA/mRNA expression from polyps and cancer in the blood. Furthermore, the study will analyze the microbiome of the intestines to explore potential associations between the gut microbiota and polyps/cancer, as well as their respective microRNA/mRNA profiles.

Primary Research Questions

Are there specific microRNA/mRNA expressions in different types of polyps/cancer and at different stages of development?

Does microRNA/mRNA expression in polyps/cancer correlate with microRNA/mRNA in the patient's blood?

Secondary Research Question Does the intestinal microbiota correlate with the presence of polyps and cancer, and their microRNA/mRNA expression?

Background Colorectal cancer is the third most frequent cancer and the second most frequent cause of cancer related death world-wide. Polyps are precursor lesions to colorectal cancer, and the transition from polyps to cancer involves the accumulation of various epigenetic and genetic changes, which is described to take approximately 10-15 years. Screening for colorectal cancer is essential, as it has been shown to reduce both morbidity and mortality. However, current screening modalities, including colonoscopy and faecal occult blood tests are challenging because of low compliance. There is currently no blood-based screening test for colorectal cancer and polyps. Understanding microRNA, non-coding RNA molecules, has opened up the possibility of developing such a test. MicroRNA, with its regulatory role in gene expression, could serve as a biomarker in the blood for colorectal polyps and cancer.

Project Description Design: Clinical Trial. The study plans to recruit 400 patients over approximately 24-48 months. The aim is to analyze microRNA/mRNA from biopsies taken from polyps, cancer, surrounding intestinal mucosa and healthy controls, and to trace these in the patient's blood. Additionally, the study will analyze the microbiota from the intestinal biopsies to investigate its role in the expression of various microRNA/mRNA. A pilot study will analyze samples from 5-20 patients, and an interim analysis will occur after including 50-100 patients. Patients over 18 years referred for colonoscopy will be asked to participate in the study

Inclusion:

Patients with colorectal polyps (approximately 150 patients). Patients with colorectal cancer (approximately 150 patients). Healthy controls with no mucosal changes during colonoscopy (approximately 100 patients).

Ethical Considerations Participation is not directly beneficial to included patients, but the knowledge we anticipate to gain from the study will hopefully it contribute to future advancements in the treatment and diagnosis of colorectal polyps and cancer. No risks are anticipated, as intestinal biopsies and blood samples are routine procedures in healthcare.

Significance In-depth information on different microRNA/mRNA expressions in colorectal polyps and cancer is expected to provide crucial knowledge leading to new diagnostic tools, treatment alternatives, and preventive measures. The study aims to establish biomarkers for blood-based screening of colorectal polyps and cancer, potentially reducing the incidence, morbidity, and mortality of colorectal cancer. The study will also investigate the significance of the microbiota in the development of polyps and cancer, aiming to contribute valuable information for understanding colorectal cancer development and potential preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years referred for colonoscopy for examination or evaluation/removal of colorectal polyps.

Exclusion Criteria:

* Patients with a history of colorectal cancer.
* Patients not in capacity to understand the study information and give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
microRNA/mRNA expression in polyps and cancer | 6 months
  Investigate specific microRNA/mRNA expressions in different types of polyps/cancer and at different stages of development
Traceability of microRNA/mRNA expression of polyps and cancer in blood | 6 months
  Investigate whether microRNA/mRNA expression in polyps/cancer correlate with microRNA/mRNA in the patient's blood

SECONDARY OUTCOMES:
Correlation of Intestinal microbiota and microRNA/mRNA expression | 6 months
  Investigate whether the intestinal microbiota correlate with the presence of polyps and cancer, and their microRNA/mRNA expression

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Malmö, section of Surgery, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided